CLINICAL TRIAL: NCT06016985
Title: National Taiwan University of Sport
Brief Title: Effects of Caffeinated Gum on a Basketball-specific Tests in Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chih-Hui Chiu (Other)
Responsible Party: Sponsor-Investigator, Chih-Hui Chiu, Professor, National Taiwan Sport University
Organization: National Taiwan Sport University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 112-1
Record Dates: First submitted 2023-08-04; First posted 2023-08-30 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Caffeine
Keywords: Eccentric exercise; basketball

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caffeine gum (Experimental): Chewed caffeine gum containing 3 mg/kg for 10 minutes
  Interventions: Dietary Supplement: caffeine gum
- placebo (Placebo Comparator): Chewed placobo gum for 10 minutes
  Interventions: Dietary Supplement: caffeine gum

INTERVENTIONS:
Dietary Supplement: caffeine gum — This study investigated the effects of chewing 3 mg/kg of caffeinated gum on basketball free throw accuracy and basketball -specific performance.
  Other Names: plocabo gum

SUMMARY:
This study investigated the effects of chewing 3 mg/kg of caffeinated gum on basketball free throw accuracy and basketball -specific performance. Fifteen trained basketball players with at least a top 8 national ranking were recruited to be participants in this study. After 2 simulation tests to familiarize the experimental procedure, we employed a double blind, randomized crossover design to divide participants into caffeine trial (CAF) and placebo trial (PL). The CAF trial chewed caffeine gum containing 3 mg/kg for 10 minutes, whereas the PL trial chewed a placebo gum without caffeine. After 15 minutes rest, the stationary free throw shooting test, countermovement jump, t-test, 20-meter segmented dash test, squat in the flywheel device and running based anaerobic sprint test were conducted.

ELIGIBILITY:
Inclusion Criteria:

* 6 years of professional basketball training and with at least a top 8 national ranking
* 6 months of continuous training,
* 3 months of recovery from sports injuries such as strains and sprains.

Exclusion Criteria:

* Non-specialized basketball players.
* has not trained regularly for the past 6 months.
* has recovered from from a sports injury for less than 3 months, or had epilepsy, hypertension, hyperlipidemia, heart disease, arthritis, osteoporosis, brain injury, or a history of caffeine allergy.
* Subjects with previous caffeine allergy response.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
stationary free throw | 15 min after intervention
  The goal percentage of stationary free throw

SECONDARY OUTCOMES:
20-meter segmented dash | 15 min after intervention
  Test the sprinting speed
fatigue index | 15 min after intervention
  Completes six 35-meter sprints at maximum effort, with a 10-second break between each sprint. The time of completion of each sprint was recorded for subsequent analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University of Sport, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-10-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT06016985/Prot_001.pdf